CLINICAL TRIAL: NCT02841761
Title: A Single-center, Open-label, Two-treatment Study to Investigate the Effect of ACT-132577 at Steady State on the Pharmacokinetics of Midazolam and Its Metabolite 1-hydroxy Midazolam in Healthy Male Subjects
Brief Title: A Study to Investigate the Effect of ACT-132577 on the Pharmacokinetics of Midazolam and 1-hydroxy Midazolam in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AC-080-103
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — aprocitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Midazolam) (Experimental): Single dose of Midazolam 8 mg on Day 1
  Interventions: Drug: Midalozam
- Treatment B1 (ACT-132577) (Experimental): Single dose of ACT-132577 150 mg on Day 2; single dose of ACT-132577 50 mg on Day 3, Day 4, and Day 5.
  Interventions: Drug: Aprocitentan
- Treatment B2 (Midazolam + ACT-132577) (Experimental): Single dose of Midazolam 8 mg and single dose of ACT-132577 50 mg on Day 6
  Interventions: Drug: Midalozam; Drug: Aprocitentan

INTERVENTIONS:
Drug: Midalozam — Syrup for oral use
  Arms: Treatment A (Midazolam); Treatment B2 (Midazolam + ACT-132577)
Drug: Aprocitentan — Capsules for oral use
  Other Names: ACT-132577
  Arms: Treatment B1 (ACT-132577); Treatment B2 (Midazolam + ACT-132577)

SUMMARY:
The purpose of this study is to evaluate the effect of ACT-132577 on the pharmacokinetics of midazolam and 1-hydroxy midazolam and to evaluate the safety and tolerability of ACT-132577 when administered alone and in combination with midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure
* Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) at screening
* Healthy on the basis of medical history, physical examination, cardiovascular assessments and serology and laboratory tests

Exclusion Criteria:

* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-01; Primary Completion 2016-09-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plama concentration (Cmax) | Midazolam PK sampling on Days 1, 2, 6 and 7
  Cmax of midazolam and 1-hydroxy midazolam following administration of midazolam alone and in combination with ACT-132577
Area under the plasma concentration-time curve from zero to infinity (AUC0-∞) | Midazolam PK sampling on Days 1, 2, 6 and 7
  AUC0-∞ of midazolam and 1-hydroxy midazolam following administration of midazolam alone and in combination with ACT-132577
Time to reach Cmax (tmax) | Midazolam PK sampling on Days 1, 2, 6 and 7
  Tmax of midazolam and 1-hydroxy midazolam following administration of midazolam alone and in combination with ACT-132577
Terminal half-life (t1/2) | Midazolam PK sampling on Days 1, 2, 6 and 7
  T1/2 of midazolam and 1-hydroxy midazolam following administration of midazolam alone and in combination with ACT-132577

SECONDARY OUTCOMES:
Number of subjects with adverse events | From Day 1 to Follow-up (for up to 38 days)
Number of subjects with serious adverse events | From Screening to Follow-up (for up to 59 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Investigator Site, Newark, New Jersey, United States